CLINICAL TRIAL: NCT01948154
Title: The Relationship of Speech Function and Quality of Life in Children With Cerebral Palsy: A Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG3C1241
Record Dates: First submitted 2013-09-05; First posted 2013-09-23 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy; Speech Function; Quality of Life
Keywords: Cerebral Palsy; Early Intervention; Speech Function; Quality of Life
MeSH Terms: conditions — Cerebral Palsy; Speech

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- children with CP: Cerebral palsy (CP) encompass a group of non-progressive, non-contagious motor conditions that cause physical disability in human development. 2-12 years old (n=60-80)
- normal child: normal child 2-12 years old (50 subjects)

SUMMARY:
Cerebral palsy (CP) encompass a group of non-progressive, non-contagious motor conditions that cause physical disability in human development. It is not infrequently to note concurrent impairment in sensory, intelligence, vision and auditory in those patients. Many studies have documented Cerebral palsy is associated with a variety of neuromotor disorders that frequently affect the speech production system. The speech function impairment varied widely due to different severity of diseases involved. The investigators hypothesize such impairment of speech function may affect degree of social participation and eventually the quality of life (QoL).

DETAILED DESCRIPTION:
Cerebral palsy (CP) encompass a group of non-progressive, non-contagious motor conditions that cause physical disability in human development. It is not infrequently to note concurrent impairment in sensory, intelligence, vision and auditory in those patients. Many studies have documented Cerebral palsy is associated with a variety of neuromotor disorders that frequently affect the speech production system. The speech function impairment varied widely due to different severity of diseases involved. The investigators hypothesize such impairment of speech function may affect degree of social participation and eventually the quality of life (QoL).

The investigators study aim in this project include: (1) to find the differences in speech function in normal developed children and in children with CP with different severity; (2) the relationship between speech function and QoL in children with CP; (3) to seek the predictable factor involving motor speech function in children with CP from the framework of International Classification of Functioning, Disability and Health - Children and Youth Version (ICF-CY).

This will be a 3-year longitudinal project recruiting 110-130 children in total. The investigators will have children with CP (n=60~80) and normal (n=50) from 2-12 years old under consent of their family. The investigator's study will be based on structure of ICF-CY. In the first year, basic clinical assessments including motor, mental, vocabulary, motor speech function, general development, and subjective questionnaires on adaptation, participation, development and quality of life will be collected. During the second to the third year, all measurements will be repeated in the end of 6- and 12-month to follow the performance of children with CP and those with normal development.

The anticipated outcomes of this study are: (1) to observe the longitudinal change of speech function and QoL in children with CP. (2) Using ICF-CY items in rehabilitation services to describe the speech function and participation of social life for children with CP. (3)To identify the influencing factors and predictors of motor speech function for children with CP.

ELIGIBILITY:
1. Subjects (Patients selection): A.50 healthy subjects B.30-40 2-5y11m y/o CP subjects C.30-40 6-12 CP subjects (children with cerebral palsy)

Inclusion Criteria:

Inclusion Criteria:

1. Parents or guardians who signed informed consent
2. Age 6-12 year old
3. Diagnosed to have cerebral palsy

Exclusion Criteria:

1. Concurrent medical condition (such as: seizure, infection)
2. Surgery within 3 months
3. Botulinum toxin-A injection within 3 months
4. Concurrent progressive or degenerative diseases, peripheral neuropathy, spinal cord injury.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will have children with CP (n=60~80) and normal (n=50) from 2-12 years old under consent of their family.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
change in General Developmental Assessment (CDIIT) in 6 month and 12 month follow up | baseline, 6 month, 12 month
  change of CDIIT

SECONDARY OUTCOMES:
change of Mental Ability | baseline, 6 month, 12 month
  change of Mental Ability (BSID-II, WPPSI-R, WISC-IV)in 6 month, 12 month follow up

OTHER OUTCOMES:
change of Motor Speech in 6 month, 12 month | baseline, 6 month,12 month
  Motor Speech Assessment (VMPAC, PCC)in 6 month, 12 month follow up
Language Assessment | baseline, 6 month, 12 month
  Language Assessment (PPVT-R; CLST)in 6 month, 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Katie P Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan